CLINICAL TRIAL: NCT06343896
Title: Evaluation of Sedation Depth and Reliability with Integrated Pulmonary Index (EPI) Follow-up in Pediatric Radiological Interventions with Effective Sedoanalgesia with BIS
Brief Title: Evaluation of Sedation Depth and Reliability with Integrated Pulmonary Index (IPI) Follow-up in Pediatric Radiological Interventions
Acronym: IPI
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: AnkaraCHBilkent-tntaygurt
Record Dates: First submitted 2024-03-27; First posted 2024-04-03 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Sedation; BIS; Integrated Pulmonary Index
Keywords: Integrated Pulmonary Index; sedoanalgesia; pediatric patient

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PEDIATRIC PATIENTS BETWEEN 2-18 YEARS OF AGE: monitorization reliability evaluation of the use of the integral pulmonary index in the child patient group
  Interventions: Other: monitorization reliability

INTERVENTIONS:
Other: monitorization reliability — evaluation of the use of the integral pulmonary index in the child patient group

SUMMARY:
In this study, we aimed to investigate the predictability of possible respiratory complications and the effect of the addition of the integrated pulmonary (EPI) score to the evaluation of the patient's respiratory index status in addition to the SPO2 measurement available in standard ASA monitoring in pediatric patients undergoing interventional radiological procedures under sedoanesthesia.

DETAILED DESCRIPTION:
This study is a single-center observational study. Patients who will undergo interventional radiologic procedures under sedoanalgesia by the radiology clinic in the pediatric operating room of the hospital will be included in the study.

This study is planned to include ASA 1-3 83 children aged 2-18 years. After obtaining the voluntary consent of the patients, anesthesia methods routinely applied in the hospital pediatric operating room will be applied.

Noninvasive blood pressure, pulse oximetry, ECG, EPI and BS monitoring will be performed. Then 4 lt/min oxygen will be started with nasal EPI cannula. Pre-processing, 0.min, 1.min, 2.min, 4.min, 6.min, 8.min,10.dk and later systolic-diastolic and average arterial blood pressure, pulse, SPO2, BIS value, EPI value, number of breaths, ETCO2 will be recorded every 5 minutes.

Apnea attacks will be recorded with ETCO2 tracking during the procedure. The capnographic criterion for an apnea episode is the inability to measure ETCO2 over a period of 15 seconds. Any apnea episode detected by clinical observation or any decrease of IPI ≤ 6 points, as well as a decrease of peripheral oxygen saturation to 92% and below, will be evaluated as hypoxia and result in an intervention including.

1. Stimulation of the patient
2. Discontinuation of the drug
3. Chin lift or chin push maneuver
4. Enhancing oxygen supplementation The necessary interventions will be performed in apnea and hypoxia states and the interventions applied when the hemodynamics of the patient is stable will be recorded The compilation time will be recorded by checking the eye opening, oral response and orientation improvement as cognitive parameters.

ELIGIBILITY:
Inclusion Criteria:

* ASA(American Society of Anesthesiologists classification) 1-2-3 ,2-18 years of age children patients who will be treated by interventional radiology

Exclusion Criteria:

* patients whose parents do not wish to participate in the research
* patients with ASA scoring greater than 4 and 4'
* Patients who are allergic to any of the drugs used or who have any contraindications for the use of the drug
* Patients with advanced organ failure (heart, kidney, liver, lung)
* Patients with intracranial mass (CIBAS), epilepsy or neuromuscular disease

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 2-18 years of age children patients who will be treated by interventional radiology
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
EVALUATION OF IPI RELIABILITY IN PEDIATRIC PATIENTS | Just before induction, 1.-2.-4.- 6.- 8-10.-15.-20.-25.-30. minutes and then every 5 minutes until the patient comes out of anesthesia. maximum duration of anesthesia was determined as 60 minutes.
  RESPIRATORY STATUS OF THE PATIENT WILL BE MEASURED BY IPI MONITOR DURING INTERVENTIONAL RADIOLOGICAL PROCEDURES PERFORMED IN PEDIATRIC PATIENTS UNDER SEDOANALGESIA

SECONDARY OUTCOMES:
BİS correlation with the IPI | Just before induction, 1.-2.-4.- 6.- 8-10.-15.-20.-25.-30. minutes and then every 5 minutes until the patient comes out of anesthesia. maximum duration of anesthesia was determined as 60 minutes.
  The researchers aim to show the effect of BIS value differences on IPI score.
pulse oximetry correlation with the IPI | Just before induction, 1.-2.-4.- 6.- 8-10.-15.-20.-25.-30. minutes and then every 5 minutes until the patient comes out of anesthesia. maximum duration of anesthesia was determined as 60 minutes.
  The researchers aim to show the effect of pulse oximetry value differences on IPI score.
noninvasive blood pressure | Just before induction, 1.-2.-4.- 6.- 8-10.-15.-20.-25.-30. minutes and then every 5 minutes until the patient comes out of anesthesia. maximum duration of anesthesia was determined as 60 minutes.
  investigators will intermittently record the intraoperative patient's noninvasive blood pressure
heart rate | Just before induction, 1.-2.-4.- 6.- 8-10.-15.-20.-25.-30. minutes and then every 5 minutes until the patient comes out of anesthesia. maximum duration of anesthesia was determined as 60 minutes.
  investigators will intermittently record the intraoperative patient's heart rate with ECG monitoring
respiratory rate | Just before induction, 1.-2.-4.- 6.- 8-10.-15.-20.-25.-30. minutes and then every 5 minutes until the patient comes out of anesthesia. maximum duration of anesthesia was determined as 60 minutes.
  investigators will intermittently record the intraoperative patient's respiratory rate
end tidal carbondioxide | Just before induction, 1.-2.-4.- 6.- 8-10.-15.-20.-25.-30. minutes and then every 5 minutes until the patient comes out of anesthesia. maximum duration of anesthesia was determined as 60 minutes.
  investigators will intermittently record the intraoperative patient's end tidal carbon dioxide value
apnea and hypoxia conditions that develop in the patient during anesthesia | Just before induction, 1.-2.-4.- 6.- 8-10.-15.-20.-25.-30. minutes and then every 5 minutes until the patient comes out of anesthesia. maximum duration of anesthesia was determined as 60 minutes.
  The investigators will record the apnea and hypoxia that develop in the patient during anesthesia and whether they are intervened or not. hypoxia will be defined as a spo2 value of 92 and below.
postoperative recovery time | the first 30 minutes in the postoperative recovery unit will be evaluated
  From the end of the operation until the patient is recovered, the patient will be followed up in the recovery unit
intraoperative total dose of medication used | at the end of the operation
  The investigators will record the total intraoperative drug dose at the end of the operation.
postoperative nausea and vomiting | the first 30 minutes in the postoperative recovery unit will be evaluated
  will be evaluated in the recovery unit within the first 30 minutes in the perioperative period.

CONTACTS AND LOCATIONS:
Overall Officials: levent ozturk, Study Chair — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Bilkent, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nelson O, Bailey PD Jr. Pediatric Anesthesia Considerations for Interventional Radiology. Anesthesiol Clin. 2017 Dec;35(4):701-714. doi: 10.1016/j.anclin.2017.08.003. PMID 29101959
- [Background] Riphaus A, Wehrmann T, Kronshage T, Geist C, Pox CP, Heringlake S, Schmiegel W, Beitz A, Meining A, Muller M, von Delius S. Clinical value of the Integrated Pulmonary Index(R) during sedation for interventional upper GI-endoscopy: A randomized, prospective tri-center study. Dig Liver Dis. 2017 Jan;49(1):45-49. doi: 10.1016/j.dld.2016.08.124. Epub 2016 Sep 1. PMID 27671621